CLINICAL TRIAL: NCT01189955
Title: The Use of Harmonic Scalpel Versus Knot Tying for Total Thyroidectomy: A Prospective Randomized Study
Brief Title: the Use of Harmonic Scalpel Versus Knot Tying for Total Thyroidectomy
Acronym: HS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Mansoura University, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: harmonic total thyroidectomy
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-02

CONDITIONS: Thyroid Swelling
Keywords: thyroidectomy; harmonic; RLN
MeSH Terms: interventions — gene 11 protein, Rotavirus B

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HS total thyroidectomy (Active Comparator): In the HS group, using the new harmonic scalpel device Focus (Ethicon Endo Surgery, Cincinnati, OH, USA) was used for cutting and coagulation . For closure of and division of superior and inferior arteries and veins we set the instrument at a power 2 i.e. more coagulation. And when smaller vessels like capsule veins we set it to the level 5 i.e. more cutting The superior artery and vein was divided close to the gland to avoid damage to superior laryngeal nerve. And control of any bleeding from the bed using the active blade of harmonic. Finally we insert drain.
  Interventions: Procedure: HS total thyroidectomy
- conventional total thyroidectomy (Active Comparator): A prophylactic antibiotic in the form of a third-generation cephalosporin was administered 2 hours before the operation. The operation was performed with the patient in the supine position under general anesthesia with endotracheal intubation. A Kocher incision, was made at the lower neck crease two finger above suprasternal notch. In the conventional group, mono- and bipolar coagulation, as well as ligatures, were allowed.
  Interventions: Procedure: conventional total thyroidectomy

INTERVENTIONS:
Procedure: HS total thyroidectomy — In the HS group, using the new harmonic scalpel device Focus (Ethicon Endo Surgery, Cincinnati, OH, USA) was used for cutting and coagulation . For closure of and division of superior and inferior arteries and veins we set the instrument at a power 2 i.e. more coagulation. And when smaller vessels like capsule veins we set it to the level 5 i.e. more cutting The superior artery and vein was divided close to the gland to avoid damage to superior laryngeal nerve. And control of any bleeding from the bed using the active blade of harmonic. Finally we insert drain.
  Other Names: Group 1
  Arms: HS total thyroidectomy
Procedure: conventional total thyroidectomy — A prophylactic antibiotic in the form of a third-generation cephalosporin was administered 2 hours before the operation. The operation was performed with the patient in the supine position under general anesthesia with endotracheal intubation. A Kocher incision, was made at the lower neck crease two finger above suprasternal notch. In the conventional group, mono- and bipolar coagulation, as well as ligatures, were allowed.
  Other Names: Group 11
  Arms: conventional total thyroidectomy

SUMMARY:
Consecutive patients treated for thyroid enlargement at our institution were evaluated for inclusion. Participants were randomly allocated to receive total thyroidectomy using harmonic scalpel HS or using ligature conventional thyroidectomy CT Follow-up visits were after 1 week, 1 month, and 6 months, Study variables included operative time, length of incision, operative bleeding, postoperative drainage, hospital stay and complication.

one hundred and thirty patients with thyroid enlargement were randomized and completed the study.

DETAILED DESCRIPTION:
Patients and method: Consecutive patients treated for thyroid enlargement at our institution were evaluated for inclusion. Participants were randomly allocated to receive total thyroidectomy using harmonic scalpel HS or using ligature conventional thyroidectomy CT Follow-up visits were after 1 week, 1 month, and 6 months, Study variables included operative time, length of incision, operative bleeding, postoperative drainage, hospital stay and complication.Preoperative preparation was performed for patients with thyrotoxicosis by antithyroid drug, and they were all euthyroid at the time of surgery. The routine pre-operative workup included measurement of thyroid-stimulating hormone and thyroid hormones (T3 and T4), as well as plasma levels of total calcium. In addition, a pre-operative laryngoscopy was performed.

A prophylactic antibiotic in the form of a third-generation cephalosporin was administered 2 hours before the operation. The operation was performed with the patient in the supine position under general anesthesia with endotracheal intubation. A Kocher incision, was made at the lower neck crease two finger above suprasternal notch.

In the HS group, using the new harmonic scalpel device Focus (Ethicon Endo Surgery, Cincinnati, OH, USA) was used for cutting and coagulation . For closure of and division of superior and inferior arteries and veins we set the instrument at a power 2 i.e. more coagulation. And when smaller vessels like capsule veins we set it to the level 5 i.e. more cutting The superior artery and vein was divided close to the gland to avoid damage to superior laryngeal nerve. And control of any bleeding from the bed using the active blade of harmonic. Finally we insert drain.

In the conventional group, mono- and bipolar coagulation, as well as ligatures, were allowed.

In both groups, the Intra-operative bleeding was estimated by weighing the gauzes before and after use. Furthermore, blood from suction (when used) was also recorded. Operation time was recorded.

Patients were discharged 24 hours after the procedure. Oral antibiotic coverage was recommended after discharge. Plasma levels of total calcium were measured on the first post-operative day. The need for oral substitution with calcium and/or vitamin D analogues during hospital stay and at patient discharge was recorded together with complications.

Follow-up was performed on postoperative day 7, and then at 1 month, 3 months, and 6 months. . Patients were also seen at our clinic if they developed symptoms between follow-up visits. At follow-up, serum thyroid hormone concentrations and serum levels of total calcium were measured, and complications recorded. Postoperative laryngoscopy was performed within 4 weeks after surgery in all patients to evaluate vocal cord function.

All assessments were conducted by investigators who were blinded to the experimental condition. The primary endpoint was operative time and secondary end points were operative bleeding, postoperative drainage, costs and complications.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients treated for thyroid enlargement

Exclusion Criteria:

* patients with one lobe pathology who need hemithyroidectomy, malignant thyroid previous neck operation, or a history of neck irradiation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
operative time | 3 hours

SECONDARY OUTCOMES:
operative bleeding | 30 days postoperative
complications | 30 days
costs | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura university, mansoura, Egypt
Locations (1):
- Ayman El Nakeeb, Mansoura, Egypt, Egypt

REFERENCES:
- [Result] Hallgrimsson P, Loven L, Westerdahl J, Bergenfelz A. Use of the harmonic scalpel versus conventional haemostatic techniques in patients with Grave disease undergoing total thyroidectomy: a prospective randomised controlled trial. Langenbecks Arch Surg. 2008 Sep;393(5):675-80. doi: 10.1007/s00423-008-0361-z. Epub 2008 Aug 2. PMID 18677509
- [Result] Siperstein AE, Berber E, Morkoyun E. The use of the harmonic scalpel vs conventional knot tying for vessel ligation in thyroid surgery. Arch Surg. 2002 Feb;137(2):137-42. doi: 10.1001/archsurg.137.2.137. PMID 11822946
- See also: mansoura university — http://www.mans.eun.eg/